CLINICAL TRIAL: NCT05335096
Title: Developing an Artificial Intelligence (AI)-Based mHealth Intervention to Improve HIV Testing in Malaysia
Brief Title: An AI-based mHealth Intervention to Improve HIV Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: University of Malaya (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2000032663; 1R21TW011663-01 (NIH); 4R33TW011663 (NIH)
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: An AI-chatbot-based mHealth intervention; Behavioral: Educational materials
- TAU group (Active Comparator)
  Interventions: Behavioral: An attention-chatbot-based mHealth intervention; Behavioral: Educational materials

INTERVENTIONS:
Behavioral: An AI-chatbot-based mHealth intervention — The participants assigned to the intervention group will get access to an AI-chatbot and can interact with the AI-chatbot at any time. In each round of the interactive communication, the chatbot will provide automated personalized messages containing PrEP, mental health, or HIV testing-related information, motivation and skills based on the participants' answers and will continuously update over time.
  Arms: Intervention group
Behavioral: An attention-chatbot-based mHealth intervention — The participants assigned to the control group will get access to an attention-chatbot and can interact with the attention-chatbot at any time. In each round of the interaction, the chatbot will provide pre-scripted time-attention health education messages to the participants.
  Arms: TAU group
Behavioral: Educational materials — the research assistant will manually sent to the participants' phone a piece of educational material and an online survey link every 30 days (at days 30, 60, 90, 120, 150 and 180).

SUMMARY:
The purpose of this study is to develop an artificial intelligence (AI)-chatbot-based mobile health (mHealth) intervention to promote HIV testing in Malaysia.

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) will be conducted in Malaysia to assess the efficacy of an AI-chatbot-based mHealth intervention versus treatment as usual (TAU) with HIV testing as the primary outcome. The primary outcome will be the proportion of participants who get tested within 180 days.

Participants will be randomized to the chatbot group and TAU group. Participants in the intervention group will get access to an AI-chatbot and can interact with the AI-chatbot at any time. In each round of the interactive communication, the chatbot will provide automated personalized messages containing pre-exposure prophylaxis (PrEP), mental health, or HIV testing-related information, motivation and skills based on the participants' answers and will continuously update over time. The participants assigned to the TAU group will get access to an attention-chatbot and can interact with the attention-chatbot at any time. In each round of the interaction, the chatbot will provide pre-scripted time-attention health education messages to the participants.

In addition to the above interventions, the research assistant will manually sent to the participants' phone a piece of educational material and an online survey link every 30 days (at days 30, 60, 90, 120, 150 and 180). The primary outcome of HIV testing will be collected through the survey.

ELIGIBILITY:
Inclusion Criteria:

* Cis-gender male
* condomless sex with men in the past 6 months
* HIV status unknown or previously tested negative
* speaks Bahasa Malaysia or English.

Exclusion Criteria:

* Does not have a smartphone
* HIV status previously tested positive
* cannot speak Bahasa Malaysia or English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 296 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants that get tested for HIV within 180 days | up to 180 days
  The number of participants who get tested for HIV within 180 days assessed by an online survey link that will be manually sent by the research assistant to the participant's phone every 30 days, up to 180 days. The survey consists of a question asking if the participant has been tested for HIV in the last 30 days with an answer of yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Ni, PhD, Principal Investigator — Yale University
Locations (1):
- University of Malaysia, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No